CLINICAL TRIAL: NCT04162704
Title: EpiCheck and Short-term Intensive Chemoresection in NMIBC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Maria Skydt Lindgren, Principal Investigator, Aarhus University Hospital
Other Study IDs: 1-10-72-207-19
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urin samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: EpiCheck — If the EpiCheck test is positive at the time of inclusion, the test is repeated prior to the fourth and sixth instillation with Mitomycin as well as prior to the subsequent two cystoscopies. If the EpiCheck test is negative at the time of inclusion, no further tests will be performed.

SUMMARY:
The aim of this explorative study is to evaluate whether EpiCheck can be used as a predictor of tumour response to short-term, intensive chemoresection with Mitomycin.

DETAILED DESCRIPTION:
The study will be conducted as an exploratory, prospective observational study. Participants consists of patients referred to short-term, intensive chemoresection due to recurrent NMIBC. The treatment adhere to the regimen described in the NICSA trial with the ClinicalTrials.gov identifier NCT03348969. Treatment consists of short-term, intensive chemoresection with Mitomycin; 40 mg is administered intravesically three times a week for two weeks. To evaluate tumour response, an early cystoscopy is performed in the outpatient clinic one to two months after treatment completion. No visible tumour and residual tumour with benign histology is considered complete response. Residual tumour tissue with neoplastic histology is considered incomplete response and will be treated with TURBT or tumour fulguration. Subsequently patients continue a standardized follow-up program as Danish guidelines prescribe which is initiated after four months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a known history of Ta HG with recurrent disease
* Patients referred to short-term, intensive chemoresection
* Patients older than 18 years

Exclusion Criteria:

* Known allergy or intolerance to Mitomycin
* Incontinence or small bladder capacity (< 100 mL)
* Previous pelvic radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a known history of Ta HG with recurrent disease and who are referred to short-term, intensive chemoresection
Sampling Method: Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
EpiCheck result | One to two months after short-term, intensive chemoresection
  Number of patients with accordance between EpiCheck score and clinical findings at the time of evaluation cystoscopy

SECONDARY OUTCOMES:
EpiCheck result 2 | One to two months after short-term, intensive chemoresection
  Number of patients with discrepancy between EpiCheck score and clinical findings at the time of cystoscopy
EpiCheck result 3 | One to two months after short-term, intensive chemoresection
  Trend of the EpiCheck test over time (increase/decrease/stable score) and its correlation to complete/incomplete tumour response
Urine cytology | One to two months after short-term, intensive chemoresection
  Sensitivity, specificity, negative and positive predictive value for urine cytology

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark